CLINICAL TRIAL: NCT04025164
Title: Hypofractionated Versus Conventional Fractionated Radiotherapy After Breast Conserving Surgery：a Multi-center Phase III Randomized Clinical Trial
Brief Title: Hypofractionated Vs Conventional Fractionated Radiotherapy After Breast Conserving Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoli Yu, Associate Professor of department of radiation oncology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-BC007
Record Dates: First submitted 2019-07-06; First posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: Hypofractionated radiotherapy; Breast Conserving Surery
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated Radiotherapy (Experimental): 40 Gy/15 fractions irradiation is delivered to the whole breast, 2.67 Gy per fraction, 5 fractions weekly.
  Tumor bed is boosted to 48 Gy simultaneously, 3.2 Gy per fraction, 5 fractions weekly.
  Interventions: Radiation: Hypofractionated Radiotherapy
- Conventional Irradiation (Active Comparator): 50 Gy/25 fractions irradiation is delivered to the whole breast, 2 Gy per fraction, 5 fractions weekly.
  Additional 10 Gy/5 fractions is boosted to tumor bed sequentially, 2 Gy per fraction, 5 fractions weekly.
  Interventions: Radiation: Conventional fractionated Radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated Radiotherapy — daily fractions, 2.66 Gy/3.2 Gy per fraction to whole breast/tumor bed, five fractions per week
  Other Names: Experimental Arm
  Arms: Hypofractionated Radiotherapy
Radiation: Conventional fractionated Radiotherapy — daily fractions, 2 Gy per fraction, five fractions per week
  Other Names: Standard Arm
  Arms: Conventional Irradiation

SUMMARY:
The study was designed to investigate whether hypofractionated radiotherapy(HF-RT) is noninferior to conventionally fractionated radiotherapy (CF-RT) in terms of tumor loco-regional control for patients after breast conserving surgery

DETAILED DESCRIPTION:
Eligible patients after breast conserving surgery will be randomized 1:1 into hypofractionated radiotherapy (HF-RT) group or conventionally fractionated radiotherapy (CF-RT) group.

Patients in HF-RT group will receive 40 Gy/15 fractions irradiation to the whole breast with/without regional lymphnodes within 3 weeks and the tumor bed is boosted to 48 Gy/15 fractions simutaneously.

Patients in CF-RT group will receive 50 Gy/ 25 fractions irradiation to whole breast with/without regional lymphnodes within 5 weeks and the tumor bed is boosted to 60 Gy/30 fractions sequentially.

The primary endpoint is loco-regional recurrence. Other cancer related events and acute/late radiation morbidities will also be evaluated. The patients will be followed for 10 years.

It is hypothesized that hypofractionated radiotherapy is non inferior to conventional fractionated radiotherapy in terms of tumor loco-regional control for patients after breast conserving surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age18-70 years
* Imaging examination confirmed single lesion. if the tumor is multiple, it needs to be removed by single quadrantectomy
* Receive breast conserving surgery with negative margins
* Axillary lymph nodes treatment: Sentinel lymph node biopsy or level I/II axillary lymph node dissection. If the sentinel lymph node is negative, the axillary lymph node dissection can be omitted. If it is positive, level I/II axillary lymph node dissection with or more than 10 lymph nodes is needed.
* The tumor bed is labeled with clips and it can be drawn on the treatment planning system.
* Pathologically confirmed invasive breast cancer
* Pathologically stage is T1-3N0-3M0
* Immunohistochemical examination is conducted to determine the status of ER, PR, HER2, Ki67 after surgery
* No distant metastases
* No supraclavicular or internal mammary nodes metastases
* No neoadjuvant chemotherapy
* Fit for postoperative radiotherapy. No contraindications to radiotherapy
* KPS≥80
* Signed informed consent

Exclusion Criteria:

* T4 or M1 breast cancer
* Supraclavicular or internal mammary nodes metastases
* Pathologically confirmed DCIS only without an invasive component
* Bilateral breast cancer or historically confirmed contralateral invasive breast cancer
* Treated with neoadjuvant chemotherapy or neoadjuvant endocrine therapy
* Multiple lesions can not be removed by single quadrantectomy
* Suspicious unresected and microcalcification, densities, or palpable abnormalities (in the ipsilateral or contralateral breast)
* KPS ≤ 70
* Patients with severe non-malignant comorbidity in cardiovascular or respiration system
* Concurrent or previous malignancy excluding basal or squamous cell carcinoma of the skin
* Previous radiotherapy to the chest wall or regional lymph node areas
* Patients with medical contraindication for radiotherapy: systemic lupus erythematosus, cirrhosis
* Pregnant or lactating
* Conditions indicating that the patient cannot go through the radiation therapy or follow up
* Unable or unwilling to sign informed consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4052 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Loco-regional recurrence (LRR) | 5 years
  Defined as any clinical and biopsy-proven tumor recurrence involving the ipsilateral chest wall and/or regional nodes (including axillary, supraclavicular, infraclavicular, or internal mammary nodes).

SECONDARY OUTCOMES:
Distant metastasis free survival (DMFS) | every 3 months during the first 2 years after the last fraction received, every 6 months during 3-5 years, every year during 6-10 years
  Distant metastasis is defined as clinical detection of metastatic disease beyond the chest wall and/or regional lymph nodes or death or last visit. Distant metastasis free survival (DMFS) is defined as the interval starting from the date of randomization until to the event.
Disease free survival (DFS) | every 3 months during the first 2 years after the last fraction received, every 6 months during 3-5 years, every year during 6-10 years
  Defined as the interval from the date of randomization to any disease recurrence or death or last visit.
Overall survival (OS) | every 3 months during the first 2 years after the last fraction received, every 6 months during 3-5 years, every year during 6-10 years
  Defined as the interval from the date of randomization to death or last visit.
Number of patients with radiation-induced acute toxicity assesses by CTCAE4.03 | before treatment, after 8 fractions (HF-RTgroup) and 15 fractions (CF-RT and HF-RT groups) and 30 fractions（CF-RT group) irradiation, 2 weeks and 3 months after the irradiation finished
  Acute toxicity (development of radiation dermatitis, pruritus, pain, radiation esophagitis, and radiation pneumonitis) will be assessed according to toxicity criteria of CTCAE version 4.03 before treatment, during treatment (after 8 fractions irradiation for HF-RTgroup and 15 fractions for CF-RT group) and the end of treatment (15 fractions irradiation for HF-RTgroup and 30 fractions for CF-RT group), 2 weeks and 3 months after the last fraction received.
Number of patients with radiation-induced late toxicity assesses by CTCAE4.03 | before treatment, every year after the last fraction received through 10 years
  Late toxicity (change of skin in irradiated area，impaired shoulder movement ，impaired shoulder movement, brachial plexopathy,ischemic heart disease) will be assessed according to toxicity criteria of CTCAE version 4.03
Number of patients with radiation-induced late toxicity assesses by LENT-SOMA Toxicity Assessment | before treatment, every year after the last fraction received through 10 years
  Development of dyspigmentation, telangiectasia in irradiated area and radiation pulmonary fibrosis will be assessed according to toxicity criteria of LENT-SOMA
Harvard/NSABP/RTOG Breast Cosmesis Grades of patients | before treatment, every year after the last fraction received through 10 years
  The cosmetic outcomes will be evaluated by radiation oncologists, nurses and patients using digital photographs and Harvard/NSABP/RTOG Breast Cosmesis Grading Scale. Harvard/NSABP/RTOG Breast Cosmesis Grading Scale classifies the overall aesthetic results in four categories from excellent, good, fair to poor.
Quality of Life Score assessed by EORTC-QLQ-C30 (version 3) | before treatment, after 15 fractions (HF-RTgroup) or 30 fractions (CF-RT group) irradiation，every year after the treatment finished through 10 years
  Patients' quality of life will be assessed using self-administered questionnaire EORTC-QLQ-C30 (version 3)
Quality of Life Score assessed by EORTC breast-cancer module (BR23) | before treatment, after 15 fractions (HF-RTgroup) or 30 fractions (CF-RT group) irradiation, every year after the last fraction received through 10 years
  Patients' quality of life will be assessed using self-administered questionnaire EORTC breast-cancer module (BR23)
Number and percentage of peripheral blood lymphocytes | before treatment, after 8 fractions (HF-RTgroup) and 15 fractions (CF-RT and HF-RT groups) and 30 fractions（CF-RT group) irradiation
  peripheral blood lymphocytes will be assessed before, during treatment (after 8 fractions irradiation for HF-RTgroup and 15 fractions for CF-RT group) and the end of treatment (15 fractions irradiation for HF-RTgroup and 30 fractions for CF-RT group). The number and percentage of peripheral blood lymphocytes will be assessed the correlation with the grade of acute toxicity assessed by CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Yu, MD, PhD, Principal Investigator — Fudan University
Locations (5):
- China (5):
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Suzhou Municipal hospital, Suzhou, Jiangsu
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Shanghai Huangpu District Central Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin K, Luo J, Yu X, Guo X. Hypofractionated radiotherapy with simultaneous tumor bed boost (Hi-RISE) in breast cancer patients receiving upfront breast-conserving surgery: study protocol for a phase III randomized controlled trial. Radiat Oncol. 2024 May 27;19(1):62. doi: 10.1186/s13014-024-02449-y. PMID 38802888